CLINICAL TRIAL: NCT05128851
Title: Prospective, Randomized, Double Blinded Trial Comparing Clinical, Radiological and Laboratory Outcomes of Hight Tibial Osteotomy With or Without Concomitant Arthroscopic Treatment of Knee Intraarticular Lesions.
Brief Title: High Tibial Osteotomy With/Without Arthroscopy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre of Postgraduate Medical Education (Other)
Responsible Party: Principal Investigator, Rafał Kamiński, Chair of Division, Centre of Postgraduate Medical Education
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: HTO_artro
Record Dates: First submitted 2020-07-03; First posted 2021-11-22 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Osteoarthritis, Knee; Meniscus; Degeneration
Keywords: HTO; Degenerative Meniscus; Osteoarthritis; Microfracture
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Fractures, Stress

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High Tibial Osteotomy and arthroscopy (Active Comparator): High Tibial Osteotomy with arthroscopically treatment of intraarticular lesions.
  Interventions: Procedure: HTO; Procedure: Arthroscopy treatment
- High Tibial Osteotomy (Sham Comparator): Descending High Tibial Osteotomy with arthroscopy without treatment of intraarticular lesions.
  Interventions: Procedure: HTO
- High Tibial Osteotomy, arthroscopy and microfractures (Active Comparator): High Tibial Osteotomy with arthroscopically treatment of intraarticular lesions and microfracture.
  Interventions: Procedure: HTO; Procedure: Arthroscopy treatment; Procedure: Micro fractures

INTERVENTIONS:
Procedure: HTO — Hight Tibial Osteotomy
Procedure: Arthroscopy treatment — Arthroscopy treatment
  Arms: High Tibial Osteotomy and arthroscopy; High Tibial Osteotomy, arthroscopy and microfractures
Procedure: Micro fractures — Micro fractures
  Arms: High Tibial Osteotomy, arthroscopy and microfractures

SUMMARY:
This study will compare Hight Tibial Osteotomy with or without arthroscopically repair intra-articular knee lesions in patients with early stages of Osteoarthritis.The purpose of this study is evaluate if addition of arthroscopy to HTO provides better clinical, radiological and laboratory outcomes.

DETAILED DESCRIPTION:
Intraarticular knee lesions are often in patients with early stages of osteoarthritis. The most frequent findings are degenerative meniscus/meniscal tears and cartilage degeneration. Degenerative meniscal lesions or meniscal tears are often incidental findings without any complains from patients. In the current literature there is no evidence for good clinical outcomes after arthroscopically treatment degenerative meniscus. Cartilage injuries are common in osteoarthritic knee and depending on grading of chondromalacia are usually treated by microfractures. By this time the choice of performed surgery depends on surgeons personal assessment. The investigators believe that concomitant intraarticular procedures added to HTO will provide better clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Knee medial compartment or patellofemoral osteoarthritis in medical interview and physical examination
* Intraarticular lesions in MRI
* Confirmation of cartilage degeneration/damage and knee malalignment in radiological tests

Exclusion Criteria:

* no informed consent to participate in the study
* age under 18 years or above 65
* multilligament injury or single plane knee instability
* another musculoskeletal disorders in lower limb
* lower limb deformity requiring axis correction below 4o or above 12.5o • joints inflammatory diseases
* ASA score > II

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-07-15 (Actual); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
KOOS | 12 months
  Knee Injury and Osteoarthritis Outcome Score
KOOS | 24 months
  Knee Injury and Osteoarthritis Outcome Score
IKDC | 12 months
  International Knee Documentation Committee - Subjective Knee Evaluation Form
IKDC | 24 months
  International Knee Documentation Committee - Subjective Knee Evaluation Form
VAS | 12 months
  Visual Analog Scale
VAS | 24 months
  Visual Analog Scale
Blood test | 2 day
  no inflammatory reaction - CRP, Il-6, CTx
Blood test | 6 weeks
  no inflammatory reaction - CRP, Il-6, CTx
Blood test | 12 weeks,
  no inflammatory reaction - CRP, Il-6, CTx

SECONDARY OUTCOMES:
Kinematic MRI with [chondrogram] | 2 day,
  Meniscus healing, cartilage quality
Kinematic MRI with [chondrogram] | 24 months
  Meniscus healing, cartilage quality
X-ray - Baldini projection | 2 day
  Patellofemoral joint measurements
X-ray - Baldini projection | 24 months
  Patellofemoral joint measurements

CONTACTS AND LOCATIONS:
Overall Officials: Rafał Kamiński, Principal Investigator — PCME, Otwock, Poland
Locations (1):
- Department of Orthopaedics and Traumatology, Centre of Postgraduate Medical Education, Professor A. Gruca Teaching Hospital, Otwock, Masovian Voivodeship, Poland